CLINICAL TRIAL: NCT06841861
Title: A Study of Therapeutic Spermatogonial Differentiation for Infertile Men Via Testicular Organoid
Brief Title: Spermatogonial Differentiation Via Testicular Organoid
Acronym: SDTO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CellARTs Inc. (Industry)
Collaborators: The Turek Clinic, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SDTO 1
Record Dates: First submitted 2024-04-26; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Infertility, Male; Gene Abnormality; Sterility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Genetic Testing; Chromosome Mapping

STUDY DESIGN:
Intervention Model Description: All participants will be donating human tissue serum (blood), skin (via biopsy), and testicular tissue (via biopsy). These samples will be used for:
  1. Primary cell culture of tissue cells will be established and genetic reprogramming could be applied to induce the long-term propagation of living cells.
  2. Characterization and genetic screening of cells will be done to discover and reveal known or novel infertility-related biomarkers or genes.
  3. Genetic reprogramming. Certain genes or gene products are inserted into donated cells to study how the cells can be changed, or reprogrammed, into embryonic-like cells or into sperm precursor cells.
  4. Culture of cells in testicular organoids. Genetically unmodified or modified cells from donated samples could be placed in a laboratory-based testicular environment to see if sperm can be made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fertile Males (Active Comparator): Fertile male participants (control group) with no known infertility conditions undergoing a vasectomy reversal. Participants will provide human tissue serum (via blood draw), skin (via biopsy), and testicular tissue (via biopsy).
  Interventions: Genetic: Stem cell; Genetic: Genetic Screening; Genetic: Genetic Reprogramming; Genetic: Cell Maturation
- Infertile Males with Genetic Sterility: Sertoli Cell Only (Experimental): Sterile male participants with unexplained or defined genetic infertility of sertoli cell only that are undergoing sperm mapping or testicular sperm retrieval (TESE) procedures. Participants will provide human tissue serum (via blood draw), skin (via biopsy), and testicular tissue (via biopsy).
  Interventions: Genetic: Stem cell; Genetic: Genetic Screening; Genetic: Genetic Reprogramming; Genetic: Cell Maturation
- Infertile Males with Genetic Sterility: Early/Late Maturation Arrest (Experimental): Sterile male participants with unexplained or defined genetic infertility of early to late maturation arrest that are undergoing sperm mapping or testicular sperm retrieval (TESE) procedures. Participant will provide human tissue serum (via blood draw), skin (via biopsy), and testicular tissue (via biopsy).
  Interventions: Genetic: Stem cell; Genetic: Genetic Screening; Genetic: Genetic Reprogramming; Genetic: Cell Maturation
- Infertile Men with Acquired Sterility (Experimental): Sterile male participants with acquired infertility from chemotherapy, infection, undecended testicles that are undergoing sperm mapping or testicular sperm retrieval (TESE) procedures. Participants will provide human tissue serum (via blood draw), skin (via biopsy), and testicular tissue (via biopsy).
  Interventions: Genetic: Stem cell; Genetic: Genetic Screening; Genetic: Genetic Reprogramming; Genetic: Cell Maturation

INTERVENTIONS:
Genetic: Stem cell — Primary cell cultures of tissue cells will be established. Cell cultures will undergo genetic reprogramming to induce the long-term propagation of living cells.
Genetic: Genetic Screening — Serum samples are processed through RNA sequencing to reveal known and novel infertility-related biomarkers and genes.
  Other Names: genome mapping; genome characterization
Genetic: Genetic Reprogramming — Genes or gene products will be reinserted into cells to observe how the cells can be changed, or reprogrammed, into embryonic-like cells or into sperm precursor cells.
Genetic: Cell Maturation — Genetically unmodified and modified cells are placed in a laboratory-based testicular environment to promote spermatogenesis into maturity.

SUMMARY:
Purpose:

This clinical trial aims to explore the potential for human sperm production in vitro by sustaining a laboratory-cultured adult testicular environment. It also seeks to identify genetic factors contributing to human sterility and failed spermatogenesis. The study's primary objectives include:

1. Identifying genomic markers associated with sterility and failed spermatogenesis.
2. Developing an ex vivo (outside the body) testis "organ-on-a-chip" ("iTestis") to support stem cell cultivation.
3. Determining whether human spermatogenesis can be re-created in vitro using stem cells nurtured in the iTestis model.

Study Description:

Researchers will analyze the genomic profiles of fertile and sterile male participants to map genetic abnormalities associated with sterility. Using testicular and skin tissue samples from participants, spermatogonial stem cells and pluripotent stem cells will be isolated and utilized to construct the ex vivo iTestis. This system will integrate genomic insights and prior research to foster human spermatogenesis outside the body.

Participant Involvement:

Participants will provide the following samples:

* Blood sample for serum analysis.
* A skin tissue biopsy.
* Testicular tissue, obtained through fine needle aspiration (FNA) or testicular sperm extraction (TESE), as part of a routine procedure.

All procedures will be conducted by the principal investigator and qualified research staff, ensuring participant safety and adherence to ethical guidelines.

ELIGIBILITY:
Inclusion Criteria: Group 1 (Fertile Control)

* Male sex of reproductive age (between 18 - 60 years old).
* Evidence of fertility or normal spermatogenesis.
* Will undergo study procedures in conjunction with their planned fertility or infertility procedures performed for clinical purposes.

Inclusion Criteria: Group 2 and 3 (Infertile)

* Male sex of reproductive age (between 18 - 60 years old).
* Males with evidence of >1 year of infertility.
* Posesses diagnosis of azoospermia is on clinical evaluation.
* Will undergo study procedures in conjunction with their planned fertility or infertility procedures performed for clinical purposes.

Exclusion Criteria:

- The lack of diagnosis of fertility or infertility, and lack of testicles.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Successful derivation of patient-specific human spermatogonial stem cells (hSSCs) from testicular tissue samples. | From initial sample collection to 24 months post all subject sample collection completion
  Metric: The presence of viable hSSCs characterized by specific molecular and cellular markers (e.g., GFRα1, PLZF) within a predefined timeframe post-derivation.
  Assessment Method: Flow cytometry, immunohistochemistry, or RT-PCR to confirm marker expression.

OTHER OUTCOMES:
Development and functional validation of an ex vivo testis organ-on-a-chip ('iTestis') platform for the cultivation and maintenance of isolated spermatogonial stem cells (hSSCs) | From the date of the first successful derivation of patient-specific hSSCs until an ex vivo testis platform is developed and can functionally cultivate and maintain the isolated spermatogonial stem cells (hSSCs), assessed for up to 24 months.
  Metric: Successful development of a biomimetic iTestis capable of maintaining hSSCs in a viable and undifferentiated state over a predefined culture period.
  Assessment Method:
  Viability: Measured by live/dead assays or metabolic activity (e.g., MTT or ATP assays).
  Stemness: Expression of hSSC markers (e.g., GFRα1, PLZF) using immunofluorescence or qRT-PCR.
Promotion of human spermatogenesis in vitro ('iSperm') using hSSCs and hiPSCs within the iTestis platform. | From the date of the initial development of the ex vivo testis platform until the promotion of human spermatogenesis using hSSCs and hiPSCs is achieved within the iTestis platform, assessed for up to 24 months.
  Metric: Generation of haploid spermatogenic cells (e.g., spermatocytes, spermatids, or sperm-like cells) from hSSCs and/or hiPSCs cultured within the iTestis platform.
  Assessment Method:
  Flow cytometry or fluorescence-activated cell sorting (FACS) to confirm haploid cell production (e.g., 1N DNA content).
  Gene and protein expression analysis of spermatogenic markers (e.g., SCP3, acrosin, protamine 1) using RT-PCR and immunofluorescence.
Successful derivation of patient-specific induced pluripotent stem cells (hiPSCs) from skin samples. | From initial sample collection to 24 months post all subject sample collection completion.
  Metric: Generation of hiPSCs that exhibit hallmark pluripotency characteristics from participant skin fibroblasts.
  Assessment Method:
  Morphological Analysis: Observation of colony morphology consistent with hiPSCs.
  Molecular and Functional Validation:
  Expression of key pluripotency markers (e.g., OCT4, SOX2, NANOG) verified by immunofluorescence, qRT-PCR, or flow cytometry.
  Functional pluripotency confirmed via in vitro differentiation into the three germ layers (endoderm, mesoderm, ectoderm).

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turek, MD, Principal Investigator — Chief Medical Officer
Locations (1):
- The Turek Clinic, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramathal C, Durruthy-Durruthy J, Sukhwani M, Arakaki JE, Turek PJ, Orwig KE, Reijo Pera RA. Fate of iPSCs derived from azoospermic and fertile men following xenotransplantation to murine seminiferous tubules. Cell Rep. 2014 May 22;7(4):1284-97. doi: 10.1016/j.celrep.2014.03.067. Epub 2014 May 1. PMID 24794432
- [Background] Kee K, Pera RA, Turek PJ. Testicular germline stem cells. Nat Rev Urol. 2010 Feb;7(2):94-100. doi: 10.1038/nrurol.2009.263. Epub 2010 Jan 19. PMID 20084076
- [Background] Kossack N, Meneses J, Shefi S, Nguyen HN, Chavez S, Nicholas C, Gromoll J, Turek PJ, Reijo-Pera RA. Isolation and characterization of pluripotent human spermatogonial stem cell-derived cells. Stem Cells. 2009 Jan;27(1):138-49. doi: 10.1634/stemcells.2008-0439. PMID 18927477
- [Background] Walsh TJ, Pera RR, Turek PJ. The genetics of male infertility. Semin Reprod Med. 2009 Mar;27(2):124-36. doi: 10.1055/s-0029-1202301. Epub 2009 Feb 26. PMID 19247914
- [Background] Durruthy-Durruthy J, Briggs SF, Awe J, Ramathal CY, Karumbayaram S, Lee PC, Heidmann JD, Clark A, Karakikes I, Loh KM, Wu JC, Hoffman AR, Byrne J, Reijo Pera RA, Sebastiano V. Rapid and efficient conversion of integration-free human induced pluripotent stem cells to GMP-grade culture conditions. PLoS One. 2014 Apr 9;9(4):e94231. doi: 10.1371/journal.pone.0094231. eCollection 2014. PMID 24718618
- [Background] Kogut I, McCarthy SM, Pavlova M, Astling DP, Chen X, Jakimenko A, Jones KL, Getahun A, Cambier JC, Pasmooij AMG, Jonkman MF, Roop DR, Bilousova G. High-efficiency RNA-based reprogramming of human primary fibroblasts. Nat Commun. 2018 Feb 21;9(1):745. doi: 10.1038/s41467-018-03190-3. PMID 29467427
- [Background] Durruthy JD, Sebastiano V. Derivation of GMP-compliant integration-free hiPSCs using modified mRNAs. Methods Mol Biol. 2015;1283:31-42. doi: 10.1007/7651_2014_124. PMID 25304205
- [Background] Huang P, Zhu J, Liu Y, Liu G, Zhang R, Li D, Pei D, Zhu P. Identification of New Transcription Factors that Can Promote Pluripotent Reprogramming. Stem Cell Rev Rep. 2021 Dec;17(6):2223-2234. doi: 10.1007/s12015-021-10220-z. Epub 2021 Aug 26. PMID 34448118
- [Background] Gaur M, Ramathal C, Reijo Pera RA, Turek PJ, John CM. Isolation of human testicular cells and co-culture with embryonic stem cells. Reproduction. 2018 Feb;155(2):153-166. doi: 10.1530/REP-17-0346. PMID 29326135
- [Background] Chui K, Trivedi A, Cheng CY, Cherbavaz DB, Dazin PF, Huynh AL, Mitchell JB, Rabinovich GA, Noble-Haeusslein LJ, John CM. Characterization and functionality of proliferative human Sertoli cells. Cell Transplant. 2011;20(5):619-35. doi: 10.3727/096368910X536563. Epub 2010 Nov 5. PMID 21054948
- [Background] Bouyer C, Chen P, Guven S, Demirtas TT, Nieland TJ, Padilla F, Demirci U. A Bio-Acoustic Levitational (BAL) Assembly Method for Engineering of Multilayered, 3D Brain-Like Constructs, Using Human Embryonic Stem Cell Derived Neuro-Progenitors. Adv Mater. 2016 Jan 6;28(1):161-7. doi: 10.1002/adma.201503916. Epub 2015 Nov 10. PMID 26554659
- [Background] Calamak S, Ermis M, Sun H, Islam S, Sikora M, Nguyen M, Hasirci V, Steinmetz LM, Demirci U. A Circulating Bioreactor Reprograms Cancer Cells Toward a More Mesenchymal Niche. Adv Biosyst. 2020 Feb;4(2):e1900139. doi: 10.1002/adbi.201900139. Epub 2020 Jan 14. PMID 32293132
- [Background] Ishii T, Pera RA. Creating human germ cells for unmet reproductive needs. Nat Biotechnol. 2016 May 6;34(5):470-3. doi: 10.1038/nbt.3559. No abstract available. PMID 27153270
- [Background] Ramathal C, Angulo B, Sukhwani M, Cui J, Durruthy-Durruthy J, Fang F, Schanes P, Turek PJ, Orwig KE, Reijo Pera R. DDX3Y gene rescue of a Y chromosome AZFa deletion restores germ cell formation and transcriptional programs. Sci Rep. 2015 Oct 12;5:15041. doi: 10.1038/srep15041. PMID 26456624
- [Background] Durruthy Durruthy J, Ramathal C, Sukhwani M, Fang F, Cui J, Orwig KE, Reijo Pera RA. Fate of induced pluripotent stem cells following transplantation to murine seminiferous tubules. Hum Mol Genet. 2014 Jun 15;23(12):3071-84. doi: 10.1093/hmg/ddu012. Epub 2014 Jan 20. PMID 24449759
- [Background] Medrano JV, Pera RA, Simon C. Germ cell differentiation from pluripotent cells. Semin Reprod Med. 2013 Jan;31(1):14-23. doi: 10.1055/s-0032-1331793. Epub 2013 Jan 17. PMID 23329632